CLINICAL TRIAL: NCT01882166
Title: Time-lapse Monitoring of Early Embryo Development After Ovarian Stimulation During Infertility Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: principal investigator left for another job, project leader retired
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/600
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Infertility, Female
Keywords: Fertilization in Vitro; Sperm Injections, Intracytoplasmic; Follicle Stimulating Hormone; Embryonic Development
MeSH Terms: conditions — Infertility, Female | interventions — Urofollitropin; follitropin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fostimon (Experimental): subcutaneous 150 IE Fostimon®. When leading follicles are > 17 mm ovulation will be induced by Ovitrelle® 500μg sc(hCG-injection). Ovum pick up (OPU) will be performed 32-36 hours later.
  Interventions: Drug: fostimon
- puregon (Experimental): subcutaneous 150 IE Puregon®. When leading follicles are > 17 mm ovulation will be induced by Ovitrelle® 500μg sc(hCG-injection). Ovum pick up (OPU) will be performed 32-36 hours later.
  Interventions: Drug: puregon

INTERVENTIONS:
Drug: fostimon
  Other Names: urinary FSH
  Arms: fostimon
Drug: puregon
  Other Names: recombinant FSH
  Arms: puregon

SUMMARY:
The number of children conceived by assisted reproductive technology is increasing in Nordic countries as well as worldwide. An important factor of success in treatment of infertility is a short "time to pregnancy" with impact on both economical aspects for the society and medical and psychological aspects for the couple. During treatment, success relies on 1) optimal stimulation of growth and maturation of multiple follicles by administration of exogenous follicle stimulating hormone (FSH), and 2) selection of the fertilized egg / embryo with the highest potential of implantation to be transferred to the mother. In the present project stimulation of egg production by human urine derived FSH (Fostimon®) and recombinant FSH (Puregon®) will be compared. To this end early embryo development and kinetics after fertilization will be evaluated. The system to be used is time-lapse recording of embryo morphology during the first days of embryo development by means of an embryoscope. Aim of this study is to investigate if Puregon and urinary Fostimon have different effect on embryo quality. The hypothesis of the study is that stimulation of egg production by these two types of follicle stimulating hormone does not have the same effect on early embryo quality.

ELIGIBILITY:
Inclusion Criteria:

* First or second intracytoplasmic sperm injection (ICSI) treatment
* BMI 18-32 kg/m²
* No previous ovarian hyperstimulation syndrome (OHSS)
* Regular menstrual cycle (cycle length 28 ± 3 days
* Less than 20 antral follicles evaluated by vaginal ultrasound
* S- Anti-Müller Hormone (AMH) 10 - 40 pmol/L
* has given informed consent

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Embryo quality | 2 days
  time-lapse recordings for all embryos will be evaluated by use of the EmbryoViewer (software developed for the EmbryoScope)

CONTACTS AND LOCATIONS:
Overall Officials: Arne Sunde, phd, Study Chair — St. Olavs Hospital
Locations (1):
- IVF Unit, St. Olavs Hospital, Trondheim, Norway